CLINICAL TRIAL: NCT07034625
Title: Comparative Evaluation of Hyaluronic Acid Spray and Low-Level Laser Therapy on Wound Healing Following Gingivectomy: A Randomized, Noninferiority Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, İpek Özgü, Dr., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AkdenizU1
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-06

CONDITIONS: Gingival Enlargement
Keywords: low-level laser therapy; gingivectomy; hyaluronic acid
MeSH Terms: conditions — Gingival Hyperplasia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low level laser therapy (Active Comparator): After gingivectomy surgery, 940 nm wavelength diode laser was applied to the wound area on the surgery day, 3rd, 5th and 7th days postoperatively. The power of the laser was set to 3W, power density 1.07 W/cm2, probe spot size 2.8 cm2, application mode continuous wave, application distance 1mm and application type stable.
  Interventions: Other: Low Level Laser Therapy
- Hyaluronic Acid Spray (Active Comparator): After gingivectomy surgery, patients were given a high molecular weight hyaluronic acid spray and instructions for use were explained. Accordingly, the patients applied the spray to the wound area twice a day for the first 7 days.
  Interventions: Other: Gengigel Spray

INTERVENTIONS:
Other: Low Level Laser Therapy — 940 nm wavelength diode laser was applied to the wound area on the surgery day, 3rd, 5th and 7th days postoperatively. The power of the laser was set to 3W, power density 1.07 W/cm2, probe spot size 2.8 cm2, application mode continuous wave, application distance 1mm and application type stable.
  Arms: Low level laser therapy
Other: Gengigel Spray — Patients were given a high molecular weight hyaluronic acid spray and instructions for use were explained. Accordingly, the patients applied the spray to the wound area twice a day for the first 7 days.
  Arms: Hyaluronic Acid Spray

SUMMARY:
Gingival enlargement is a common condition caused by increased cell numbers, leading to connective tissue expansion. It can hinder plaque control and cause aesthetic and functional problems, often requiring surgical intervention. Gingivectomy is the primary procedure for treating gingival enlargement, ensuring periodontal health. Postoperative low-level laser therapy (LLLT) may reduce inflammation, relieve pain, and accelerate tissue regeneration. Similarly, hyaluronic acid (HA) stimulates cell proliferation, migration, and differentiation, promoting wound healing. This study aimed to compare the effects of LLLT and HA spray on early wound healing after gingivectomy.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* Having chronic inflammatory gingival hyperplasia affecting at least 6 teeth symmetrically in the maxillary or mandibular anterior region with gingivectomy indication
* No usage of any medication affecting periodontal tissues or causing gingival hyperplasia such as antiepileptics, immunosupresors or calcium channel blockers
* No history of periodontitis with attachment and bone loss

Exclusion Criteria:

* Having systemic disease
* Pregnancy or breastfeeding
* Smoking
* Inadequate oral hygiene
* Antibiotic usage for the past six months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score | 2 weeks
  The Visual Analogue Scale (VAS) is the most common method used to translate values that we cannot measure numerically into numerical form and to measure the severity of acute pain; therefore, the pain felt by the patients in the postoperative period was evaluated using VAS. Patients were given a chart in which a line with a length of 10 cm and a number between 1 and 10 was written on each cm distance and the definitions of the parameter to be evaluated were written and the patient was asked to indicate where his/her condition was appropriate on this line by pointing. On the given scale, 'no pain' was written on '0' end and 'worst pain' was written on the '10' (0: No pain 1-3: Slight pain 3.1-6: Moderate pain 6.1-10: Severe pain), and the patient was asked to mark his/her current pain condition on this line on the 1st day, 3rd day, 7th day and 14th day after the operation.
Wound Healing Area Assessment | 2 weeks
  At baseline, 3rd day, 7th day and 14th day, the surgical gingivectomy area was disclosed by a erythrosin and gluten-free plaque-disclosing solution to visualize the areas in which the gingival epithelium is absent, abraded or lacking sufficient keratinization and to distinguish these areas from normal gingiva.

SECONDARY OUTCOMES:
Gingival Index | 6 weeks
  The GI was measured at six sites per tooth, according to Löe & Silness:
  0- Normal gingiva;
  1. Mild inflammation with slight color change, mild alteration of gingival surface structure and no bleeding on probing;
  2. Moderate inflammation with edema, redness, swelling and bleeding on probing;
  3. Severe inflammation with marked edema and redness, ulceration and tendency to bleed spontaneously.
Full Mouth Bleeding Score | 6 weeks
  FMBS: BoP index is taken as present/absent (+/-) at six sites/teeth, full mouth bleeding score (FMBS) was then calculated as a percentage.
Probing Pocket Depth | 6 weeks
  Probing pocket depth were taken at six sites/tooth and recorded using a Williams periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Nezahat Arzu Kayar, PhD, DDS, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Uslu MO, Akgul S. Evaluation of the effects of photobiomodulation therapy and ozone applications after gingivectomy and gingivoplasty on postoperative pain and patients' oral health-related quality of life. Lasers Med Sci. 2020 Sep;35(7):1637-1647. doi: 10.1007/s10103-020-03037-8. Epub 2020 May 20. PMID 32435906
- [Background] Reddy SP, Koduganti RR, Panthula VR, Surya Prasanna J, Gireddy H, Dasari R, Ambati M, Chandra G B. Efficacy of Low-level Laser Therapy, Hyaluronic Acid Gel, and Herbal Gel as Adjunctive Tools in Gingivectomy Wound Healing: A Randomized Comparative Clinical and Histological Study. Cureus. 2019 Dec 21;11(12):e6438. doi: 10.7759/cureus.6438. PMID 31993275
- [Background] Ozcelik O, Cenk Haytac M, Kunin A, Seydaoglu G. Improved wound healing by low-level laser irradiation after gingivectomy operations: a controlled clinical pilot study. J Clin Periodontol. 2008 Mar;35(3):250-4. doi: 10.1111/j.1600-051X.2007.01194.x. PMID 18269665
- [Background] Yakout BK, Kamel FR, Khadr MAEA, Heikal LAH, El-Kimary GI. Efficacy of hyaluronic acid gel and photobiomodulation therapy on wound healing after surgical gingivectomy: a randomized controlled clinical trial. BMC Oral Health. 2023 Oct 27;23(1):805. doi: 10.1186/s12903-023-03519-5. PMID 37891549